CLINICAL TRIAL: NCT06697548
Title: Conservative Care for Pelvic Pain (C2P2) in Women Service Members: A Multisite, Multigroup Non-inferiority Randomized Clinical Trial With Development of Clinical Decision Tools
Brief Title: Conservative Care for Pelvic Pain (C2P2) in Women Service Members
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR230127; HT94252410709 (Other Grant/Funding Number: Department of Defense (DoD))
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pelvic Pain
Keywords: Pelvic health; Chronic pelvic pain; Physical therapy; Military; womens health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Usual Care Group will receive their current medical management care along with study-specific patient education and progressive home exercise.
  Interventions: Other: Lumbopelvic and Hip Therapeutic Exercise; Other: Chronic Pelvic Pain Education
- Emerging Field-expedient Care (Experimental): Emerging Field-expedient Care Group will receive a combination of emerging nonvaginal interventions aimed at normalizing sensory, motor, and autonomic nervous system dysfunction including pain neuroscience education, diaphragmatic breathing training, and lumbopelvic manual therapy and dry needing treatment
  Interventions: Other: Pain Neuroscience Education; Other: Lumbopelvic and Hip Therapeutic Exercise; Other: Extrapelvic Manual Therapy; Other: Extrapelvic Dry Needling; Other: Deep Paced Diaphragmatic Breathing Training; Other: Chronic Pelvic Pain Education
- Gold-standard Intravaginal Specialist Care (Active Comparator): Gold-standard Intravaginal Specialist Care Group will receive tailored intravaginal and intrarectal manual therapy and biofeedback intervention by a pelvic-health specialist.
  Interventions: Other: Pain Neuroscience Education; Other: Lumbopelvic and Hip Therapeutic Exercise; Other: Deep Paced Diaphragmatic Breathing Training; Other: Chronic Pelvic Pain Education; Other: Intravaginal and intrarectal pelvic floor physical therapy

INTERVENTIONS:
Other: Pain Neuroscience Education — Participants will watch and discuss a short (5-minute) standardized pain neuroscience education video with their treating provider. The video explains and illustrates how chronic pain is different than acute pain in that it concerns nervous system hypersensitivity more than local tissue damage. Pain neuroscience education principles from the video will then be used to throughout all interventions to coach the participants through graded exposure of activities that may have previously been painful or provoked anxiety.
  Arms: Emerging Field-expedient Care; Gold-standard Intravaginal Specialist Care
Other: Lumbopelvic and Hip Therapeutic Exercise — These motor control exercises will focus on proprioception, coordination, and sensorimotor control training and include progressive exercises that focus on transversus abdominis, lumbar multifidus, diaphragmatic, pelvic floor muscles, and deep hip stabilizers. Exercises will progress from more stabilized (e.g., pelvic tilt, cat and cow) to less stabilized and more dynamic and functional (e.g., forward bending, eccentric squat) to mimic the demands of work duty. Exercise will be trained and progressed during the clinical visits and be performed daily at home.
Other: Extrapelvic Manual Therapy — Thrust and non-thrust manual therapy will be applied to the lumbar facet, sacroiliac, and hip joints based upon the clinical exam in a semi-standardized manner
  Arms: Emerging Field-expedient Care
Other: Extrapelvic Dry Needling — Dry needling treatment to muscles of the lumbopelvic and upper thigh regions in a semi-standardized manner based upon a palpatory examination. The palpatory examination will include the erector spinae, lumbar multifidi, gluteus medius/minimus, piriformis, illiacus, and hip adductor muscles.
  Arms: Emerging Field-expedient Care
Other: Deep Paced Diaphragmatic Breathing Training — The breathing intervention will start with education describing the link between the diaphragm and the pelvic floor to include awareness of any breath holding patterns and finding positions that facilitate expansion of the ribs, abdominals, and pelvic floor muscles with inhalation. Then progressive training will be given to encourage deep breathing at a pace of approximately 6 breaths per minute.
  Arms: Emerging Field-expedient Care; Gold-standard Intravaginal Specialist Care
Other: Chronic Pelvic Pain Education — During the first visit, participants will receive and briefly discuss the 2023 standardized patient educational handout created by the International Pelvic Pain Society with their treating provider. The educational handout describes chronic pelvic pain etiology, typical symptoms, examination, and treatments.
Other: Intravaginal and intrarectal pelvic floor physical therapy — Superficial vulvar, perineal and intravaginal manual therapy and biofeedback utilizing commonly used techniques in previous research selected based on identified impairments from the pelvic floor examination will be performed.
  Arms: Gold-standard Intravaginal Specialist Care

SUMMARY:
This study will test the effectiveness of emerging conservative interventions for treatment of chronic pelvic pain (CPP) that can be performed without intravaginal specialization. Participants with CPP will be randomly assigned to one of three groups. The first group will receive treatment based on what they normally would receive, including medications, education, and exercise (Usual Care Group). The second group will receive contemporary non-vaginal treatment including manual therapy, dry needling, and specific breathing training (Emerging Field-expedient Care Group). The third group will receive intravaginal treatment by a pelvic health specialist (Gold-standard Intravaginal Specialist Care Group). Participants will be asked about their pain and symptoms and have measurements taken of their pelvic and back muscles after 1, 3, 6, and 12 months. In addition to seeing which treatments work best, clinical decision tools (using medical and trauma history along with clinical examination) will be developed to identify women with CPP likely to respond favorably to non-vaginal conservative interventions. This study will help determine the best non-vaginal treatment strategies for women with CPP and help clinicians quickly determine which patients are likely to benefit from treatment by non-pelvic health physical therapists (e.g., in theater), vs. patients who should be referred for pelvic health specialty care.

DETAILED DESCRIPTION:
This trial will measure both clinical outcomes (pain, pelvic floor symptoms, work/duty absenteeism) and physiologic outcomes (pelvic floor and lumbopelvic muscle function and pain sensitivity) at 1 week and after 1, 3, 6, and 12 months of three different conservative physical therapy treatments. It is hypothesized that women who receive emerging field-expedient care will report greater improvements than those who receive only usual care, and their outcomes will be no worse than women who receive gold-standard intravaginal specialist care. Additionally, clinical decision tools incorporating characteristics from medical and trauma history, along with clinical examination, will be developed to identify women with CPP likely to respond favorably to emerging field-expedient care vs. requiring gold-standard intravaginal specialist care.

ELIGIBILITY:
Inclusion Criteria:

1. Pain of at least 3 months duration in the abdominal-lumbopelvic area, defined as below the umbilicus, between the two ilia, and above the pubic symphysis including the vulvar, perineal, and vaginal regions.

Exclusion Criteria:

1. Sign that pelvic pain may be due to other serious medical issue (recent history of abdominal pelvic surgery, current infection, disrupted tissue integrity, neoplasm, or history of radiation to the pelvic floor tissue or the tissues being measured for stiffness).
2. Chronic debilitating medical conditions (e.g., fibromyalgia, lupus, complex regional pain syndrome, multiple sclerosis or other progressive neurologic condition).
3. Currently pregnant or pregnancy in the last 6 months.
4. Body mass index over 33 (Waco participants only due to limitation of the instrumentation).
5. Soldiers in an Advanced Individual Training (AIT) status.
6. Previous intervention to address lumbopelvic muscle stiffness or pain such as dry needling, injections, or soft tissue intervention of any kind in the past 6 months.
7. Inability to read English at an 8th grade reading level (any participant unable to read the informed consent form, which will be written at an 8th grade level).
8. Inability to legally provide informed consent for any other reason.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The Pelvic Floor Distress Inventory (PFDI-20) | 1 week and 1, 3, 6, and 12 months
  The Pelvic Floor Distress Inventory (PFDI-20) is a 20-item questionnaire that assesses the frequency and severity of pelvic floor symptoms. It consists of 3 subscales: the pelvic floor distress inventory 6 (POPDI-6), the colorectal anal distress inventory 8 (CRADI-8), and the urinary distress inventory 6 (UDI-6). Each question is rated on a scale of 0-4 with 0 representing "no symptoms," and 4 representing "quite a bit." Higher scores represent more bothersome symptoms.
The Genitourinary Pain Index (GUPI) | 1 week and 1, 3, 6, and 12 months
  The Genitourinary Pain Index (GUPI) is 9-item questionnaire that assesses presence, location, frequency, quality and quantity of genitourinary pain in both men and women.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS) | 1 week and 1, 3, 6, and 12 months
  Participants will rate their current pain on a scale of 0-10 with zero being no pain at all and 10 being the worst pain imaginable. Subjects will also rate their worst pain within the past week and their pain at its best within the last week, to gain an assessment of variability and intensity of pain.
Pelvic Floor Muscle Tone | 1 week and 1, 3, 6, and 12 months
  On a subset of 150 participants, pelvic floor muscle tone will be estimated from shear wave elastography ultrasound (US).
Superficial Lumbopelvic Muscle Tone | 1 week and 1, 3, 6, and 12 months
  On a subset of 150 participants, resting tone of several lumbopelvic muscles will be measures using a MyotonPRO device.
Pelvic Floor Pain Sensitivity | 1 week and 1, 3, 6, and 12 months
  On a subset of 150 participants, pelvic floor pain sensitivity will be assessed using pain algometry.
Lumbopelvic Muscle Pain Sensitivity | 1 week and 1, 3, 6, and 12 months
  On a subset of 150 participants, Pain sensitivity of the same lumbopelvic muscles and locations assessed using the MyotonPRO will be measured using a digital hand-held pressure algometer.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - U.S. Army Medical Center of Excellence (MEDCoE), San Antonio, Texas
  - Baylor University, Waco, Texas

IPD SHARING:
Plan to Share IPD: No
Depending upon where the findings of this study are published, sharing individual participant data might not be feasible.